CLINICAL TRIAL: NCT01450124
Title: Safety, Tolerability And Mechanism Of Action Of Boswellic Acids In Multiple Sclerosis and Clinically Isolated Syndrome: A MRI-Controlled, Multicenter, Baseline-To-Treatment, 32-Weeks, Open-Label, Phase IIa Trial
Brief Title: Safety, Tolerability And Mechanism Of Action Of Boswellic Acids (BA) In Multiple Sclerosis (SABA)
Acronym: SABA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: inims-03
Record Dates: First submitted 2011-09-18; First posted 2011-10-12 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boswellic acids (BOSWELAN) (Experimental): Baseline to treatment single arm - 4 months baseline and 8 months of treatment at a t.i.d. (Ter In Die (Latin: Three Times A Day) dose of between 400-1600 mg of BOSWELAN.
  Interventions: Drug: Boswellic acids (BOSWELAN)

INTERVENTIONS:
Drug: Boswellic acids (BOSWELAN) — 8 months of treatment at a t.i.d. (Ter In Die (Latin: Three Times A Day) dose of between 400-1600 mg Boswelan
  Other Names: BOSWELAN

SUMMARY:
To determine the safety and tolerability of BOSWELAN in subjects with multiple sclerosis or clinically isolated syndrome and to describe the effect of Boswellic acids on the disease activity as assessed by monthly MRI measures.

DETAILED DESCRIPTION:
Boswellic acids (BAs), the main biologically active compound of frankincense, are orally available and known to exhibit anti-inflammatory activities. This is a Phase IIa bicentric baseline-to-treatment study with the standardized frankincense extract Boswelan to test the safety, tolerability and efficacy of BAs in RR-MS patients. Following a 3-month screening phase, patients received an individualized dose finding identifying the highest well tolerated BOSWELAN dose for each patient. The primary outcome in the treatment phase (Stage 3) will first compare mean Gd-enhancing lesion number occurring during the 4 month baseline to mean Gd-enhancing lesion number occurring months 5, 6, 7, 8 on treatment in patients treated with a dose of at least 800 mg t.i.d.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years, inclusive*
* Females and Males (as no specific gender-related differences are expected, no specific gender distribution is planned. See GCP-V § 7 (2) Nr. 12)
* Subjects with a clinically isolated syndrome (high risk of conversion to MS) as well as subjects with clinically definite relapsing-remitting according to published criteria (50)
* Diseases with similar clinical neurological symptoms (e.g. lues, borreliosis, collagenosis or vasculitis) have been excluded by differential diagnostics
* EDSS score between 0.0 and 5.5, inclusive.
* Baseline MRI Lesion frequency of 0.5 or greater
* Patients are clinically stable, i.e. without relapse and not having received steroids within 30 days prior to inclusion
* Patients have either failed standard treatment (interferon beta, glatiramer acetate) by clinical measures or were not eligible for any of the standard treatments available or opted not to start or to continue with any of these treatments

Exclusion Criteria:

* ALT (SGPT) or AST (SGOT) > three times the upper limit of normal
* Total white blood cell count < 3,000/mm3
* Platelet count < 85,000/mm3
* Creatinine > 1.5 mg/dl
* Serology indicating active hepatitis B or C infection or other chronic liver disease
* Positive pregnancy test, or breast-feeding female
* Nausea/vomiting as a frequent complaint
* History or signs of immunodeficiency
* Concurrent, clinically significant (as determined by the investigator) cardiac, immunological, pulmonary, neurological, renal, and/or other major disease

If prior treatment was received, the subject must have been off treatment for the required period prior to enrollment (see Table 2).

Table 2: Restrictions on pre-treatments Agent Glatiramer acetate (CopaxoneTM), Interferon beta (BetaferonTM, AvonexTM, RebifTM) IV Ig, Azathioprine (ImurekTM), Methotrexate, Cyclophosphamide (CytoxanTM), Mitoxantrone, plasma exchange, Cyclosporine, oral myelin, Cladribine, natalizumab, and other immunosuppressive treatments Corticosteroids, ACTH Time required off agent prior to enrollment 12 weeks 24 weeks 8 weeks Prior treatment with any other investigational drug or procedure for MS will be evaluated individually by the investigators.

* History of alcohol or drug abuse within the 5 years prior to enrollment
* Female subjects who are not post-menopausal or surgically sterile who are not using an highly effective method of birth control. Highly effective is defined as having a failure rate of <1%.

Written documentation that the subject is post- menopausal or surgically sterile must be available prior to study start

* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's returning for follow-up visits on schedule
* Previous participation in this study
* Participation in other pharmaceutical trials during this study or 3 months before
* Patients hospitalized due to juridical or legal regulation
* Known hypersensitivity to BA
* Known contraindications for MRI examinations including hypersensitivity to gadolinium, severe renal insufficiency, a mechanical heart valve or any kind of metallic implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean number of total Gd-enhancing lesions | 8 months
  Mean number of Gd-enhencing lesions comparing a baseline/pre-treatment interval of 3 months to a 3 months interval on treatment

SECONDARY OUTCOMES:
Number of new active lesions (new Gd-enhancing lesions +new or enlarging non-enhancing T2 lesions) | 8 months
Relapse rate | 8 months
  Annualized Relapse rate - comparing baseline to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - NeuroCure Clinical Research Center (NCRC), Berlin
  - University Medical Centre Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Derived] Faizy TD, Broocks G, Thaler C, Rauch G, Gebert P, Sturner KH, Flottmann F, Leischner H, Kniep HC, Stellmann JP, Heesen C, Fiehler J, Gellissen S, Hanning U. Development of Cortical Lesion Volumes on Double Inversion Recovery MRI in Patients With Relapse-Onset Multiple Sclerosis. Front Neurol. 2019 Feb 22;10:133. doi: 10.3389/fneur.2019.00133. eCollection 2019. PMID 30873106